CLINICAL TRIAL: NCT04378491
Title: Tro_Le_Tomy - Clinical and Functional Outcome After Lateral Trochlear Lengthening Osteotomy
Brief Title: Clinical and Functional Outcome After Lateral Trochlear Lengthening Osteotomy Lateral Trochlear Lengthening Osteotomy
Acronym: Tro_Le_Tomy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01405; ch20Muendermann2
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Patellar Instability
Keywords: lengthening osteotomy of the lateral trochlea; Lateral trochlear lengthening osteotomy; trochlear dysplasia Dejour type A or B; short lateral articular trochlea
MeSH Terms: interventions — Muscle Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of clinical measurements — Collection of clinical measurements:
  * Active and passive range of motion (ROM) of the knee, hip and ankle Joint bilaterally.
  * Passive patellar translation in 30° of flexion billaterally in quadrants of translation.
  * Patellar apprehension test (Fairbank's Test) and the Moving Patellar Apprehension (MPAT) test for the diagnosis of patellar instability. The Fairbank's Test is performed in 30° of Flexion while the MPAT is performed while flexing the knee from 0° to 90°.
Other: Collection of data for muscle strength — Collection of data for muscle strength:
  * Muscle strength will be measured bilaterally using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA). For the knee, maximum isokinetic Flexion and extension torques will be collected between full extension and full flexion at a movement speed of 60°/s (3 x 5 repetitions) Maximum joint torques in each movement direction will be recorded for each joint and normalized to body weight
Other: Collection of EMG Data — Collection of EMG Data:
  * Surface electrodes will be placed bilaterally on the vastus medialis and lateralis rectus femoris, biceps femoris and semitendinosus muscles following the guidelines of the SENIAM project (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles). Simultaneously with the muscle strength measurements, EMG data will be collected using a 12-channel EMG system (myon AG, Schwarzenberg, Switzerland, sampling rate 2400 Hz).
Other: Collection of Clinical Scores — Collection of Clinical Scores:
  * patient's pain, range of motion and ability to perform daily living activities will be assessed using the Kujala Anterior Knee Pain Scale, Lysholm Knee Score, visual analog scale score (VAS) and the Tegner Activity Score
Other: Collection of Imaging Data - Radiological measurements — Collection of Imaging Data - Radiological measurements: Xrays and MRIs which were already performed as part of the original diagnostic and follow-up procedures pre- and postoperative will be reviewed and analysed.

SUMMARY:
The purpose of this study is to evaluate the functional and clinical outcome of this new lengthening osteotomy of the lateral trochlea in patients with patella instability, trochlear dysplasia Dejour type A or B, short lateral articular trochlea quantified by the lateral condyle index and presence of a lateral trochlear bump.

DETAILED DESCRIPTION:
A short lateral articular trochlea leads to failure in stabilizing the patella close to full Extension of the knee. To address this type of pathology, a trochlear lengthening osteotomy was described. To date only case reports describing the clinical outcome of this new osteotomy exist and information on functional outcome regarding muscle strength and electromyography (EMG) data is lacking. The purpose of this study is to evaluate the functional and clinical outcome of this new lengthening osteotomy of the lateral trochlea in patients with patella instability, trochlear dysplasia Dejour type A or B, short lateral articular trochlea quantified by the lateral condyle index and presence of a lateral trochlear bump.

ELIGIBILITY:
Inclusion Criteria:

* 2 years (as of September 2019) since conducting a lateral trochlear lengthening osteotomy

Exclusion Criteria:

* Inability to provide informed consent
* Neurological disorders potentially affecting lower extremity muscle strength.
* Surgery involving the patellofemoral joint prior to the lateral trochlear lengthening osteotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated between 01/2014 and 09/2017 (n=6) with lateral trochlear lengthening osteotomy at the Clinic of Orthopaedics and Traumatology at the University Hospital Basel
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
presence of a recurrent patellar dislocation/ radiological reduction of the trochlear bump postoperative by plain radiograph of the knee/ lateral view | at Baseline
  presence of a recurrent patellar dislocation postoperative by plain radiograph of the knee/ lateral view:
  * crossing sign: The sign is positive when the trochlear groove lies in same plane as anterior border of lateral condyle. It represents a flattened trochlear groove
  * double contour sign: The sign is positive when the anterior border of lateral condyle lies anterior to anterior border of medial condyle. It represents a convex trochlear groove/hypoplastic medial condyle
  * presence of a lateral trochlear bump prominence
  * the patellar height will be evaluated according to Insall-Salvati method (normal between 0.8 and 1.2) and Caton Deschamps method (normal between 0.6 and 1.3)
presence of a recurrent patellar dislocation/ radiological reduction of the trochlear bump postoperative by Skyline patellar view | at Baseline
  The trochlea form will be assessed, the existence of trochlear dysplasia will be confirmed and classified according to Dejour
(Change in) Lateral condyle index assessed by MRI of the knee | at Baseline
  Lateral condyle index assessed by MRI of the knee (preoperative (always conducted) and in the cases where they are available postoperative MRIs). The lateral condyle index was designed to measure the lateral trochlea by comparing the anterior cartilaginous trochlea (a) and the posterior aspect (p) [(a:p)× 100].

SECONDARY OUTCOMES:
Subjective Evaluation of the outcome of the operation | at Baseline
  The patients will be asked to subjectively evaluate the outcome of the operation according to the following options:
  * Excellent: Patient is fully recovered and has resumed all activity without restrictions
  * Somewhat Improved: Patient is mostly recovered and has resumed a majority of activities
  * Unchanged: Patient outcome is equivalent to pre-operative complaints
  * Somewhat Worse: Patient is experiencing symptoms worse than pre-operative complaints
  * Significantly Worse: Patient outcome is worse than pre-operative complaints with significantly worse symptoms
Kujala Anterior Knee Pain Scale (AKPS) | at Baseline
  The Kujala AKPS is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. For example, a 'Limp' score would be scored as follows: none (5), slight/periodic (3), constant (0). Total scores range from 0 to 100.
Lysholm Knee Score | at Baseline
  The Lysholm Knee Score consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions, and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disability.
Visual analog scale score (VAS) | at Baseline
  The visual analogue scale (VAS) is a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable.
Tegner activity scale | at Baseline
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.

CONTACTS AND LOCATIONS:
Overall Officials: +41 (0)61 32 87133 Muendermann, Prof., Principal Investigator — Orthopädie/Traumatologie, University Hospital Basel
Locations (1):
- Orthopädie/Traumatologie, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Ismailidis P, Egloff C, Nuesch C, Mundermann A, Pagenstert G. Lateral trochlear lengthening osteotomy. Arch Orthop Trauma Surg. 2021 Oct;141(10):1721-1730. doi: 10.1007/s00402-020-03736-5. Epub 2021 Feb 24. PMID 33625541